CLINICAL TRIAL: NCT05661643
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of Temozolomide in Advanced Gastrointestinal Stromal Tumor Patients With SDH Deficiency
Brief Title: The Efficacy and Safety of Temozolomide in SDH-deficient GIST
Acronym: GIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2203
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- temozolomide treatment (Experimental)
  Interventions: Drug: Temozolomide capsule

INTERVENTIONS:
Drug: Temozolomide capsule — Temozolomide 200 mg/m2 is administered orally for 1-5 days of each cycle, and then canceled for 23 days (a total of 28 days is 1 cycle)

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of temozolomide in SDH deficiency GIST patients.

DETAILED DESCRIPTION:
Wild type GISTs are less responsive to imatinib with a response rate of 23.1-44.6% and a median progressiion-free survival of 12.3-12.8 months. The efficacy of imatinib is limited in particular in SDH deficienctGIST with a reported response of 2%. Therefore, the development of a new therapeutic agents is urgently needed.

Recently, a study of TKI-resistant SDH-deficient preclinical model showed that temozolomide, an alkylating agent, promotes DNA damage in tumor cells, leading to tumor cell killing. In a retrospective analysis, 2 out of 5 SDH deficient GIST patients treated with temozolomide showed partial response, suggesting its efficacy in this patient population.

Based on these findings,The goal of this clinical trial is to investigate the efficacy and safety of temozolomide in SDH deficiency GIST patients. In addition, for exploratory purposes, aim to investigate the efficacy and safety of temozolomide in KIT and PDGFRA wild-type GIST without SDH deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 years or older, at the time of acquisition of informed consent
2. Histologically confirmed GIST with CD117(+), DOG-1(+)
3. Wild type GIST without KIT or PDGFRα gene mutations determined by Sanger sequencing and panel sequencing
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 ~ 2
5. Resolution of all adverse events with prior treatments to grade 0 or 1 by NCI-CTCAE version 5.0
6. At least one measurable lesion by RECIST version 1.1.
7. Adequate bone marrow, hepatic, renal, and other organ functions, before adjuvant imatinib treatment

   * Neutrophil >1,500/mm3
   * Platelet > 100,000/mm3
   * Hemoglobin >8.0 g/dL
   * Total bilirubin < 1.5 x upper limit of normal (ULN)
   * AST/ALT < 2.5 x ULN
   * Creatinine <1.5 x ULN
8. Life expectancy ≥12 weeks
9. Disease progression or discontinuation of treatment due to intolerable toxicity at least with palliative 1st line imatinib .
10. Washout period of previous TKIs or chemotherapy for more than 4 times the half life ((Imitinib and regorafenib need 1 week and sunitinib need 2 weeks.)
11. Provision of a signed written informed consent

Exclusion Criteria:

1. Confirmed GIST with KIT or PDGFRα gene mutations determined by Sanger sequencing and panel sequencing
2. Women of child-bearing potential who are pregnant or breast feeding
3. Women or men who are not willing to use effective contraception entering the study period or until at least 6 months after the last study drug administration
4. If any of the following applies within ≤ 6 months prior to starting study enrollment : Myocardial Infarction, severe instable angina, coronary/peripheral bypass, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack, treatment required severe arrhythmia
5. Uncontrolled infection
6. Acute and chronic liver disease and all chronic liver impairment.(But Patients with stable chronic hepatitis B are eligible
7. Acute, or chronic medical or psychiatric condition or laboratory abnormality such as active uncontrolled infection that difficult to study participation in the judgment of the investigator
8. Known diagnosis of HIV infection (HIV testing is not mandatory).
9. History of another primary malignancy that is currently clinically significant or currently requires active intervention.
10. Alcohol or substance abuse disorder
11. The patients with NTRK fusion

5)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective respone rate in SDH deficiency wild type GIST | up to 4 years
  complet response+partial response defined by RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea